CLINICAL TRIAL: NCT02421952
Title: Clinical Use of Baxter Animated Retching Faces (BARF) Scale in Children
Acronym: BARF
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mary Felberg, Pediatric Anesthesiologist, Baylor College of Medicine
Other Study IDs: H32386
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Cohort: All subjects will be asked to assess their pain and nausea using the visual analogue scales (VAS), the modified faces scale and the BARF scale as described below in the preoperative and postoperative areas.

SUMMARY:
Pediatric research in the management of nausea has been limited by the absence of a reliable method to quantify the intensity of this subjective symptom. In adults, the visual analog scale (VAS) is an accurate tool, but this has not been shown to be reliable in young children. By default the most common objective outcome measure used in pediatric studies has been the incidence and number of emetic episodes. This measure, however, correlates poorly with the somatic subjective symptom of nausea.

DETAILED DESCRIPTION:
Pediatric research in the management of nausea has been limited by the absence of a reliable method to quantify the intensity of this subjective symptom. In adults, the visual analog scale (VAS) is an accurate tool, but this has not been shown to be reliable in young children. By default the most common objective outcome measure used in pediatric studies has been the incidence and number of emetic episodes. This measure, however, correlates poorly with the somatic subjective symptom of nausea.

Apfel et al have shown that 30-40% of adult patients undergoing surgery have post discharge nausea and / or vomiting while 12% have vomiting. These data on nausea in adults were based on a visual analog scale for nausea. There are no data on the incidence of postoperative nausea in children since the severity of symptoms are difficult to measure as younger children are known to be unable to use the VAS reliably.

Recently a pictorial scale for measuring nausea, the Baxter Animated Retching Faces (BARF) scale, has been developed and shown to have construct, content and convergent validity as an instrument to measure nausea in children. The clinical usefulness of this scale in determining the incidence of postoperative and post-discharge nausea in children has yet to be determined including the lowest age where it can be used reliably, the score associated with a patient's perception of a need for treatment, the minimum change in the scores of clinical relevance and the test-retest reliability when nausea is rated as not having changed.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 3 years but below 18 years
2. Elective surgery
3. American Society of Anesthesiologists physical status 1-3 (Free from major concurrent disorders)
4. Free from nausea and / or vomiting in the previous 24 hours
5. Cognitive, visual, hearing and communicative ability to use the VAS as shown by the ability to complete a seriation task in which children pick the biggest of 6 cut out shapes, then the smallest, and the biggest remaining until no shapes remain (Beyer et al: J Pediatr Nurs 1992; 7: 335-46)

Exclusion Criteria:

1. Developmental delay
2. Blindness
3. Impaired cognitive or communicative abilities including inability to rate the intensity of symptoms and failure to complete the seriation task
4. Surgical procedures which may result in diminished hearing or vision in the immediate postoperative period
5. Nausea and /or vomiting within 24 hours prior to the procedure
6. Inability to understand English,
7. Patient or parental refusal to participate
8. Pregnant females

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pre-operative patients at Texas Children's Hospital
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2013-04; Primary Completion 2018-03-08 (Actual); Study Completion 2018-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Felberg, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watcha MF, Lee AD, Medellin E, Felberg MT, Bidani SA. Clinical Use of the Pictorial Baxter Retching Faces Scale for the Measurement of Postoperative Nausea in Children. Anesth Analg. 2019 Jun;128(6):1249-1255. doi: 10.1213/ANE.0000000000003850. PMID 31094795

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Cohort: The study design is a cross sectional study of patients undergoing surgery. There was no group assignment, no placebo group and each subject was his or her own control. All patients were asked to assess their pain and nausea using the visual analogue scales (VAS), the modified faces scale, and the BARF scale in the preoperative and postoperative areas.
Period: Overall Study
Arm/Group | Single Cohort
Started | 208
Excluded From PACU and Post-Analysis (Reasons itemized below) | 16
Included in PACU Analysis | 192
Completed (Diary returned) | 99
Not Completed | 109
Not completed — Diary Not Returned | 93
Not completed — Failed seriation task | 13
Not completed — Subject uncooperative for baseline test | 2
Not completed — Surgery cancelled | 1

BASELINE CHARACTERISTICS:
Population: 208 subjects screened for the ability to use VAS and Pictorial Scales. 16 subjects excluded from PACU and Post-discharge analysis for failed seriation task, being uncooperative during baseline assessment, or having their surgery cancelled after consent was obtained.
Arm/Group | Single Cohort
Number analyzed (Participants) | 208
Age, Customized [Count of Participants; unit: Participants]
  3-3.9 years | 32
  4-4.9 years | 18
  5-5.9 years | 26
  6-6.9 years | 18
  7-7.9 years | 21
  8-11.9 years | 71
  12-17.9 years | 22
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 124
  Female | 67
  Unknown | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 208
Could use BARF for all time points [Count of Participants; unit: Participants] | 190

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Nausea, Emesis, Severe Nausea, Severe Emesis and Number Receiving Rescue Antiemetics in the Post-Anesthetic Care Unit (PACU)
Description: To measure pain and nausea, subjects completed the VAS and two pictorial scales (Faces Pain Scale-Revised for pain and BARF for nausea). The VAS uses a horizontal 10cm line with the extremes of "no pain at all" and "worst pain imaginable". The subject marks on the line their pain rating. Higher points indicate more severe or intense pain. FACES scale has 6 faces with assigned scores ranging from 0 to 10 with a score difference of 2 between each face (a higher score indicates more pain). The BARF scales has 6 faces with assigned scores ranging from 0 to 10 with a score difference of 2 between each face (a higher score indicates more nausea).
Time Frame: When awake and responding to commands in the post-anesthesia care unit (PACU)
Population: Patients with severe nausea were included in the number with any nausea. Patients with severe emesis were included in the number with any emesis. Because some patients had both nausea and vomiting, the sum of the number with nausea and the number with emesis will not equal those with either nausea or emesis.
Measure: Count of Participants; unit: Participants
Groups:
- Single Cohort: Includes subjects who consented to participate, passed the seriation task, remained cooperative during the baseline assessment, and whose surgeries were not cancelled following informed consent.
Arm/Group | Single Cohort
Number analyzed (Participants) | 192
Participants
  Any Nausea | 60
  Severe Nausea (Score >6) | 13
  Any Emesis | 8
  Severe Emesis (>= 3 episodes) | 2
  Rescue Antiemetics | 16
  Postoperative Nausea OR Vomiting | 62
  Postoperative Nausea AND Vomiting | 6

2. Secondary Outcome: Incidence of Post-Discharge Nausea, Emesis, Severe Nausea, Severe Emesis and Number Receiving Rescue Antiemetics in Subjects Who Returned the Diary
Description: Patients were discharged from the PACU when they achieved institutional discharge criteria. The parents were given a diary to record the maximum nausea on the VAS and BARF scales during the first 24 postoperative hours. Each child's caretaker was contacted by phone 24 hours after surgery to determine whether the child had any nausea or vomiting and which medications were given after discharge. The VAS uses a horizontal 10cm line with the extremes of "no pain at all" and "worst pain imaginable". The subject marks on the line their pain rating. Higher points indicate more severe or intense pain. FACES scale has 6 faces with assigned scores ranging from 0 to 10 with a score difference of 2 between each face (a higher score indicates more pain). The BARF scales has 6 faces with assigned scores ranging from 0 to 10 with a score difference of 2 between each face (a higher score indicates more nausea).
Time Frame: First 24 postoperative hours
Measure: Count of Participants; unit: Participants
Arm/Group | Single Cohort
Number analyzed (Participants) | 99
Participants
  Nausea | 34
  Severe Nausea Score >6) | 15
  Any Emesis | 16
  Severe Emesis (>= 3 episodes) | 3
  Rescue Antiemetics | 8
  Post-Discharge Nausea OR Vomiting | 39
  Post-Discharge Nausea AND Vomiting | 11

3. Secondary Outcome: Age-Related Ability to Use the BARF Scale
Description: The age-related ability to use the BARF scale was determined by constructing receiver operating characteristic (ROC) curves and calculating the area under the ROC curve and the 95% confidence interval (CI), along with sensitivity and specificity.
Time Frame: Comprehensive
Population: All enrolled subjects were included.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Sensitivity; Specificity: ROC Curve Using Age as Cutoff Points
Arm/Group | Sensitivity | Specificity
Number analyzed (Participants) | 208 | 208
percentage
  3-3.9 years | 100 [97.5 to 100] | 0 [0 to 22.9]
  4-4.9 years | 89.5 [84 to 93.3] | 70.6 [44 to 88.6]
  5-5.9 years | 81.1 [74.6 to 86.2] | 82.4 [55.8 to 95.3]
  6-6.9 years | 68.9 [61.8 to 75.3] | 100 [77.1 to 100]
  7-7.9 years | 59.5 [52.1 to 66.5] | 100 [77.1 to 100]
  8-11.9 years | 48.4 [41.2 to 55.7] | 100 [77.1 to 100]
  12-17.9 years | 11.6 [7.5 to 17.1] | 100 [77.1 to 100]

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events while active in the study (from enrollment until diaries were completed at 24 hours PACU discharge).
Description: This is a minimal risk, cross-sectional study of pain and nausea using three scales. There was no randomization or intervention.
Arm/Group | Single Cohort
All-Cause Mortality (participants affected / at risk) | 0/208
Serious Adverse Events (participants affected / at risk) | 0/208
Other Adverse Events (participants affected / at risk) | 0/208

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT02421952/Prot_SAP_000.pdf